CLINICAL TRIAL: NCT01356784
Title: Efficacy of "Tailored Physical Activity or" "Chronic Pain Self-management Program" on Returning to Work: a Randomized Controlled Trial in Sicklisted Citizens With Chronic Pain Related to the Spine or Upper Body
Brief Title: Returning to Work. Efficacy of "Tailored Physical Activity or" "Chronic Pain Self-management Program" in Sicklisted Citizens With Chronic Musculoskeletal Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: DK-Sønderborg Municipality (Unknown)
Responsible Party: Principal Investigator, Lotte Nygaard Andersen, Ph.d. fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 95-154-32028
Record Dates: First submitted 2011-05-13; First posted 2011-05-19 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Musculoskeletal Pain
Keywords: Sick-listed; Tailored physical activity; Patient education; Returning to work; DK-Sønderborg Municipality; columna; upper body
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tailored Physical Activity (Experimental)
  Interventions: Other: Tailored Physical Activity
- "Chronic Pain Self-management Programme" (Active Comparator)
  Interventions: Behavioral: "Chronic Pain Self-management Programme"
- Health Counselling (Other)
  Interventions: Behavioral: Health counselling

INTERVENTIONS:
Other: Tailored Physical Activity — Health counselling (1,5h) and graded physical activity (3×50 min/week in 10 weeks)
  Arms: Tailored Physical Activity
Behavioral: "Chronic Pain Self-management Programme" — Health counselling (1,5h) and 'Chronic Pain Self-management Program' (2,5h in 6 weeks)
  Arms: "Chronic Pain Self-management Programme"
Behavioral: Health counselling — Health guidance (1,5h)
  Arms: Health Counselling

SUMMARY:
TEst the effect of "Tailored Physical Activity" or "Chronic Pain Self-management Program" on Returning to Work in Sicklisted Citizens With Chronic Pain Related to the Spine or Upper Body

DETAILED DESCRIPTION:
Pain affects quality of life and it's important for the individual who experience chronic pain to find strategies to prevent or reduce pain. In some situations pain can't be reduced and the individual has to master pain by learning to live with it. Pain can lead to a loss of functions which may change one's roles both in relation to the family as to colleagues, for example sick leave from work.

Limited evidence is available on the effects of interventions to sick-listed citizens with chronic musculoskeletal pain.

This study test the effect of either "tailored physical activity or "Chronic Pain Self-management Program" on returning to work and the parameters pain, function and quality of life respectively on the body function and participation level of sick-listed people with chronic musculoskeletal pain related to columna and the upper body.

Citizens in DK-Sønderborg Municipality sick-listed for a maximum of 9 weeks will be invited. Participants will be randomized for either tailored physical activity, "Chronic Pain Self-Management Program" or reference group.

Primary endpoint is 3 months and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Sick-listed with musculoskeletal pain related to columna or the upper body for a maximum period of 9 weeks in DK-Sønderborg Municipality

Ages: 18 Years to 66 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sick-listed or not | 3 months
  Registration of the participants status as sick-listed or not and co-primary the number of days on sick-leave in the period.

SECONDARY OUTCOMES:
Aerobic capacity | 3 months
hand-grip strength | 3 months
Body weight, waist circumference, hip circumference | 3 months
Questionnaire | 3 months
Sick-listed or not | 12-months follow-up
  Registration of the participants status as sick-listed or not and co-primary the number of days on sick-leave in the period.
Aerobic capacity | 12-months follow-up
Hand-grip strength | 12-months follow-up
Questionnaire | 12-months follow-up
Body weight, waist circumference, hip circumference | 12 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Health Care Centre, Sønderborg, Denmark

REFERENCES:
- [Derived] Andersen LN, Juul-Kristensen B, Roessler KK, Herborg LG, Sorensen TL, Sogaard K. Efficacy of 'Tailored Physical Activity' or 'Chronic Pain Self-Management Program' on return to work for sick-listed citizens: design of a randomised controlled trial. BMC Public Health. 2013 Jan 23;13:66. doi: 10.1186/1471-2458-13-66. PMID 23343386
- See also: University of Southern Denmark — http://www.sdu.dk